CLINICAL TRIAL: NCT00128193
Title: Two New Leprosy Skin Test Antigens: MLSA-LAM and MLCwA Phase II Study in a Leprosy-Endemic Region
Brief Title: Leprosy Skin Test Antigens Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 00-002
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Results first posted 2010-11-01 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2010-08

CONDITIONS: Leprosy
Keywords: leprosy, Mycobacterium leprae, Hansen's Disease, skin test, Nepal
MeSH Terms: conditions — Leprosy | interventions — Tuberculin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- A1-Ramping (MLSA-LAM) (Experimental): 5 subjects to receive: 1.0 mcg of MLSA-LAM, 0.1 mcg of MLSA-LAM, 5 TU Purified Protein Derivative/Tubersol®, saline (NaCl).
  Interventions: Other: MLSA-LAM; Biological: Tuberculin, Purified Protein Derivative; Other: Placebo
- C1-Target Population (Experimental): 80 subjects to receive: 1.0 mcg of MLSA-LAM, 1.0 mcg of MLCwA and 2TU Purified Protein Derivative/RT-23.
  Interventions: Biological: Tuberculin, Purified Protein Derivative; Other: MLSA-LAM; Other: MLCwA
- C-1b-Target Population (Low Dose) (Experimental): 80 subjects to receive: 0.1 mcg MLSA-LAM, 0.1 mcg MLCwA, 2 TU Purified Protein Derivative/RT-23.
  Interventions: Biological: Tuberculin, Purified Protein Derivative; Other: MLSA-LAM; Other: MLCwA
- B2-Full-Scale (MLCwA) (Experimental): 45 subjects to receive: 1.0 mcg of MLCwA, 0.1 mcg of MLCwA, 5 TU Purified Protein Derivative/Tubersol®, saline (NaCl).
  Interventions: Other: MLCwA; Biological: Tuberculin, Purified Protein Derivative; Other: Placebo
- B1-Full-Scale (MLSA-LAM) (Experimental): 45 subjects to receive: 1.0 mcg of MLSA-LAM, 0.1 mcg of MLSA-LAM, 5 TU Purified Protein Derivative/Tubersol®, saline (NaCl).
  Interventions: Other: MLSA-LAM; Biological: Tuberculin, Purified Protein Derivative; Other: Placebo
- A2-Ramping (MLCwA) (Experimental): 5 subjects to receive: 1.0 mcg of MLCwA, 0.1 mcg of MLCwA, 5 TU Purified Protein Derivative/Tubersol®, saline (NaCl).
  Interventions: Other: MLCwA; Biological: Tuberculin, Purified Protein Derivative; Other: Placebo

INTERVENTIONS:
Biological: Tuberculin, Purified Protein Derivative — A tuberculin skin test used to diagnose latent tuberculosis (TB) infection. 2 TU dose
  Arms: C-1b-Target Population (Low Dose); C1-Target Population
Other: MLSA-LAM — Mycobacterium leprae soluble antigen with minimal amounts of immunosuppressive lipoglycans; dosages 0.1 and 1.0 micrograms; administered in sterile diluent 0.9% saline (NaCl).
  Arms: A1-Ramping (MLSA-LAM); B1-Full-Scale (MLSA-LAM); C-1b-Target Population (Low Dose); C1-Target Population
Other: MLCwA — Cell wall-associated proteins of Mycobacterium leprae; dosages 0.1 and 1.0 micrograms; administered in sterile diluent 0.9% saline (NaCl).
  Arms: A2-Ramping (MLCwA); B2-Full-Scale (MLCwA); C-1b-Target Population (Low Dose); C1-Target Population
Biological: Tuberculin, Purified Protein Derivative — Licensed TB reagent, 100 microliters, 5 TU dose.
  Arms: A1-Ramping (MLSA-LAM); A2-Ramping (MLCwA); B1-Full-Scale (MLSA-LAM); B2-Full-Scale (MLCwA)
Other: Placebo — Saline (NaCl) serves as a diluent control in Stage A and B only.
  Arms: A1-Ramping (MLSA-LAM); A2-Ramping (MLCwA); B1-Full-Scale (MLSA-LAM); B2-Full-Scale (MLCwA)

SUMMARY:
The purpose of this study is to see how healthy people and leprosy patients react to 2 new skin tests for detecting leprosy. The study will evaluate the new skin tests that may aid in measuring the number of people exposed to leprosy and enable its diagnosis and treatment at an earlier stage. Participant's ages 18-60 living in Kathmandu, Nepal will be enrolled. Stages A and B of the study will use the skin test in healthy volunteers. Stage C will use the skin test in high risk volunteers (including individuals with leprosy), healthy individuals in contact with leprosy patients and individuals with tuberculosis (TB, lung disease). Study procedures will include injections, physical exam, and blood testing. Injection sites will be checked several times during the participant's study involvement (5 hours of time spread over approximately 1 month). Volunteers screened for the study, which have leprosy or tuberculosis will be treated or referred for treatment.

DETAILED DESCRIPTION:
This double-blind Phase II clinical trial will be conducted in 3 stages to evaluate 2 new leprosy skin test antigens, Mycobacterium (M.) leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) and M. leprae Cell Wall Antigen (MLCwA), as diagnostic-epidemiological tools designed to measure incidence of leprosy infection in Kathmandu, Nepal, a leprosy endemic area. Stage A will provide an initial indication of safety of the 2 new test antigens in 10 healthy members of the leprosy endemic population (5 subjects per antigen at 2 dosages each). Stage B will expand this analysis by an additional 90 healthy subjects (45 subjects per antigen). If any subjects in Stage A or B show ulcerations at the 1.0 mcg dose of MLSA-LAM or MLCwA test sites, then only the 0.1 mcg dose will be used for Stage C. The final stage, Stage C, is divided into 2 parts. The first part, Stage C-1, will assess safety of both antigens at the high dose (1.0 mcg) in populations at a higher risk of developing ulcerations at skin test sites. Eighty subjects will be recruited: 20 household contacts of Borderline Lepromatous Leprosy (BL) / Lepromatous Leprosy (LL) leprosy patients, 20 BL/LL leprosy patients, 20 Borderline Tuberculoid Leprosy (BT) / Tuberculoid Leprosy (TT) patients and 20 tuberculosis (TB) patients. The second part, Stage C-1b, is a continuation of Stage C-1 with the same number of subjects recruited from the same groups to assess the reactivity of both antigens at the low dose (0.1 mcg). This study will define a positive skin test reaction for MLSA-LAM and MLCwA, and this definition will be used in estimating sensitivity and specificity for each skin test antigen and dosage. It is expected that the BT/TT leprosy patients and healthy contacts of leprosy patients will have larger indurations at both M. leprae-derived antigen sites and a variable reaction at the tuberculin/Purified Protein Derivative (PPD) site. The non-contacts, BL/LL leprosy patients, and TB patients will have smaller indurations at all leprosy skin test sites and a variable reaction at the tuberculin/PPD site. Finally, the TB patients will react with a large induration at the tuberculin/PPD site. Primary study objectives are to evaluate safety of these 2 new leprosy skin test antigens and to estimate specificity and sensitivity of these skin test antigens in detecting M. leprae infection by: selecting a dosage of the MLSA-LAM and MLCwA antigens that causes minimal induration in healthy non-exposed subjects; selecting a size of induration that will serve as a definition of a positive skin test reaction for MLSA-LAM and MLCwA in leprosy patients; and comparing proportion of positive skin test reactors in healthy subjects to proportion in BT/TT and BL/LL leprosy patients, contacts of leprosy patients, and TB patients. Secondary study objectives are to compare mean size of induration in response to each test antigen in healthy subjects versus BT/TT and BL/LL leprosy patients, contacts of leprosy patients, and TB patients as a measure of specificity and sensitivity; to compare the specificity and sensitivity of the 2 new antigens with tuberculin/PPD in patients with clinical leprosy, contacts of leprosy patients, and healthy unexposed subjects (non-patient contacts); to quantify release of IFN-gamma from lymphocytes in whole blood from leprosy patients, leprosy patient contacts, TB patients, and healthy nonexposed subjects, following in vitro stimulation with leprosy skin test antigens and PPD, using the QuantiFERON-CMI (Cellestis Limited, Valentia California) kit. Results will be compared to the magnitude of the skin test response; and to determine if antibodies against a M. leprae specific anti

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Between the ages of 18 and 60 years old
* Male or female; not less than 30 percent for one gender
* Agree to participate in the study after verbal explanation by the physician and nurses, as indicated by signing an informed consent form
* Weight greater than 30 Kg (female) and 38 Kg (male)
* Available for skin test readings
* Nepali residents, including expatriates from India

Healthy, Non-Contacts

* Healthy (determined by history and physical examination)
* No household or working contact with tuberculosis or leprosy patients

Contacts of Leprosy Patients

* Healthy (determined by history and physical examination)
* Household contact of a person with leprosy for at least 6 months duration, and within 6 months of this study, or a person professionally exposed to leprosy for at least 5 years duration, and within 6 months of this study

Persons with Leprosy

* Having one or more of the following symptoms:

  1. Hypopigmented or erythematous skin lesion(s) with definite loss of sensation
  2. Damage to the peripheral nerves as demonstrated by palpable thickening with or without impairment of sensation and/or weakness of the muscles of hands, feet or face
  3. Presence of acid-fast bacilli in slit skin smears
  4. Histological changes diagnostic of leprosy in skin biopsy
* Receiving standard multi drug treatment for leprosy or completed treatment for leprosy no more than 4 years prior to study enrollment

Persons with Tuberculosis

* Having active tuberculosis as defined by one of the following:

  1. Extra-pulmonary tuberculosis if confirmed by culture
  2. Pulmonary tuberculosis, defined as:
* Having a history of a productive cough of more than 3 weeks duration that may be accompanied by night sweats, loss of appetite, haemoptysis, weight loss, chest pain, or shortness of breath, and
* Having one or more of the following diagnostic criteria:
* Sputum smear-positive, defined as one or more of the following: at least 2 of 3 successive sputum samples positive for acid-fast bacilli by microscopy; or at least one sputum specimen positive and x-ray abnormalities consistent with pulmonary tuberculosis; or at least one positive sputum specimen that is culture positive for Mycobacterium tuberculosis
* Sputum smear-negative, defined as three sputum specimens negative for acid-fast bacilli but with x-ray evidence consistent with pulmonary tuberculosis and that does not clear with non-tuberculosis antibiotics; or three sputum samples negative for acid-fast bacilli by microscopy but culture positive for Mycobacterium tuberculosis
* Completed the intensive phase of chemotherapy for tuberculosis, but still undergoing the continuation phase of therapy

Exclusion Criteria:

All subjects

* Pregnant (as determined by a urine pregnancy test performed on females of child-bearing age on Day 0, prior to admission into the study) or lactating females
* Currently on oral corticosteroid or other immunosuppressive treatment
* Cancer, diabetes, or other chronic illness
* Extra-pulmonary tuberculosis not confirmed by culture
* Known hypersensitivities or allergies
* Expatriates other than those from India
* Participation in an earlier stage of this study
* Concurrent participation in another clinical trial

Healthy, Non-Contacts

* History of treated tuberculosis or leprosy
* Clinical signs of leprosy or tuberculosis
* Known contact with persons with leprosy or tuberculosis

Healthy Contacts of Leprosy Patients

* History of treated tuberculosis or leprosy
* Clinical signs of leprosy or tuberculosis

Persons with Leprosy

* Leprosy patients in reversal reaction or erythema nodosum leprosum (ENL) reaction or those being treated with corticosteroids or thalidomide for these conditions
* History of treated tuberculosis
* Clinical signs of tuberculosis
* Completed full course of standard multidrug treatment (MDT) for leprosy more than 4 years prior to study enrollment

Persons with Tuberculosis

* History of treated leprosy
* Clinical signs of leprosy
* Completed full course of standard tuberculosis treatment
* Known contact with leprosy patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2002-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Colorado State University - Microbiology, Immunology & Pathology, Fort Collins, Colorado, United States
- Nepal (5):
  - Anandaban Hospital, Kathmandu
  - Green Pastures Hospitals, Kathmandu
  - Lalitpur Nursing Campus, Kathmandu
  - Patan Hospital, Kathmandu
  - Tribhuvan University - Anandaban Hospital, Kathmandu

REFERENCES:
- [Result] Rivoire BL, Groathouse NA, TerLouw S, Neupane KD, Ranjit C, Sapkota BR, Khadge S, Kunwar CB, Macdonald M, Hawksworth R, Thapa MB, Hagge DA, Tibbals M, Smith C, Dube T, She D, Wolff M, Zhou E, Makhene M, Mason R, Sizemore C, Brennan PJ. Safety and efficacy assessment of two new leprosy skin test antigens: randomized double blind clinical study. PLoS Negl Trop Dis. 2014 May 29;8(5):e2811. doi: 10.1371/journal.pntd.0002811. eCollection 2014. PMID 24874401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Stage A (10) and B (90) participants were recruited from Lalitpur Nursing Campus in Kathmandu, Nepal. All participants for stages C1 (80) and C1b (80) were recruited from either Anandaban Hospital in Kathmandu, Nepal or Patan Hospital in Lalitpur, Nepal. Enrollment occurred between 30Apr2002 and 12Aug2009.
Groups:
- A1 - MLSA in Healthy Non-Exposed Participants: 5 healthy non-exposed participants received 1.0 mcg of Mycobacterium (M.) leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM), 0.1 mcg of MLSA-LAM, 5 tuberculin units (TU) Purified Protein Derivative(PPD)/Tubersol®, saline (NaCl)
- A2 - MLC in Healthy Non-Exposed Participants: 5 healthy non-exposed participants received 1.0 mcg of M. leprae Cell Wall Antigen (MLCwA), 0.1 mcg of MLCwA, 5 TU Purified Protein Derivative/Tubersol®, saline (NaCl)
- B1 - MLSA in Healthy Non-Exposed Participants: 45 healthy non-exposed participants received 1.0 mcg of MLSA-LAM, 0.1 mcg of MLSA-LAM, 5 TU Purified Protein Derivative/Tubersol®, saline (NaCl)
- B2 - MLC in Healthy Non-Exposed Participants: 45 healthy non-exposed participants received 1.0 mcg of MLCwA, 0.1 mcg of MLCwA, 5 TU Purified Protein Derivative/Tubersol®, saline (NaCl)
- C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients: 20 borderline lepromatous/lepromatous (BL/LL) leprosy patients received 1.0 mcg of MLSA-LAM, 1.0 mcg of MLCwA and 2TU Purified Protein Derivative/RT-23
- C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients: 20 borderline tuberculoid/tuberculoid (BT/TT) leprosy patients received 1.0 mcg of MLSA-LAM, 1.0 mcg of MLCwA and 2TU Purified Protein Derivative/RT-23
- C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts: 20 healthy contacts of BL/LL leprosy patients received 1.0 mcg of MLSA-LAM, 1.0 mcg of MLCwA and 2TU Purified Protein Derivative/RT-23
- CI - High Dose MLSA and MLC in TB Patients: 20 tuberculosis (TB) patients received 1.0 mcg of MLSA-LAM, 1.0 mcg of MLCwA and 2TU Purified Protein Derivative/RT-23
- C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients: 20 borderline lepromatous/lepromatous (BL/LL) leprosy patients received 0.1 mcg MLSA-LAM, 0.1 mcg MLCwA, 2 TU Purified Protein Derivative/RT-23
- C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients: 20 borderline tuberculoid/tuberculoid (BT/TT) leprosy patients received 0.1 mcg MLSA-LAM, 0.1 mcg MLCwA, 2 TU Purified Protein Derivative/RT-23.
- C1b - Low Dose MLSA and MLC in Healthy Contacts: 20 healthy contacts of BL/LL leprosy patients received 0.1 mcg MLSA-LAM, 0.1 mcg MLCwA, 2 TU Purified Protein Derivative/RT-23.
- C1b - Low Dose MLSA and MLC in TB Patients: 20 TB patients received 0.1 mcg MLSA-LAM, 0.1 mcg MLCwA, 2 TU Purified Protein Derivative/RT-23.
Period: Overall Study
Arm/Group | A1 - MLSA in Healthy Non-Exposed Participants | A2 - MLC in Healthy Non-Exposed Participants | B1 - MLSA in Healthy Non-Exposed Participants | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Started | 5 | 5 | 45 | 45 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
Completed | 5 | 5 | 42 | 44 | 18 | 17 | 16 | 20 | 18 | 18 | 17 | 18
Not Completed | 0 | 0 | 3 | 1 | 2 | 3 | 4 | 0 | 2 | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A1 - MLSA in Healthy Non-Exposed Participants | A2 - MLC in Healthy Non-Exposed Participants | B1 - MLSA in Healthy Non-Exposed Participants | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients | Total
Number analyzed (Participants) | 5 | 5 | 45 | 45 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 13 | 10 | 0 | 0 | 0 | 4 | 0 | 1 | 4 | 1 | 33
  Between 18 and 65 years | 5 | 5 | 32 | 35 | 20 | 20 | 20 | 16 | 20 | 19 | 16 | 19 | 227
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (6.4) | 29.4 (2.9) | 21.1 (5.3) | 23.1 (6.7) | 37.5 (12.3) | 32.9 (12.9) | 32.9 (11.0) | 26.0 (7.7) | 35.2 (13.1) | 39.0 (13.5) | 30.2 (12.1) | 31.1 (13.1) | 28.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 14 | 8 | 6 | 6 | 7 | 7 | 5 | 4 | 14 | 5 | 84
  Male | 1 | 1 | 31 | 37 | 14 | 14 | 13 | 13 | 15 | 16 | 6 | 15 | 176
Region of Enrollment [Number; unit: participants]
  Nepal | 5 | 5 | 45 | 45 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 260

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reactions to the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 0.1 Microgram
Description: Participants returned to the clinic at Days 2 (Group A), 3 (all groups) and 7 (Groups B and C), and at Day 28 if reactions were still present (all groups), for reader measurements of erythema and induration and assessment of other adverse events of pain/tenderness, bleeding, urticaria, infection, or blistering/ulcerating. Participants are counted if they had any measurable erythema or induration, or reported any of the other listed adverse events. Reactions were reported as present or absent, and were not graded for severity.
Time Frame: Up to 28 Days
Population: All participants who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Groups:
- A1 - MLSA in Healthy Non-Exposed Participants: 5 healthy non-exposed participants received 1.0 mcg of Mycobacterium (M.) leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM), 0.1 mcg of MLSA-LAM, 5 TU Purified Protein Derivative(PPD)/Tubersol®, saline (NaCl)
Arm/Group | A1 - MLSA in Healthy Non-Exposed Participants | B1 - MLSA in Healthy Non-Exposed Participants | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 5 | 45 | 20 | 20 | 20 | 20
Participants
  Erythema | 0 | 3 | 1 | 5 | 4 | 2
  Induration | 0 | 2 | 0 | 4 | 2 | 0
  Pain/Tenderness | 0 | 1 | 0 | 0 | 1 | 0
  Bleeding | 0 | 0 | 0 | 0 | 1 | 0
  Urticaria | 0 | 0 | 0 | 0 | 1 | 0
  Infection | 0 | 0 | 0 | 0 | 1 | 0
  Blistering/Ulcerating | 0 | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Participants With the Reaction of Itching to the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 0.1 Microgram
Description: Itching was assessed for participants in Groups B and C only, who returned to the clinic at Days 3 and 7, and at Day 28 if reactions were still present. Itching was reported as present or absent, and not graded for severity.
Time Frame: Up to 28 Days
Population: All participants in Groups B and C who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | B1 - MLSA in Healthy Non-Exposed Participants | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 45 | 20 | 20 | 20 | 20
Participants | 0 | 0 | 1 | 1 | 0

3. Primary Outcome: Number of Participants With Reactions to the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 1.0 Microgram
Description: Participants returned to the clinic at Days 2 (Group A), 3 (all groups) and 7 (Groups B and C), and at Day 28 if reactions were still present (all groups), for reader measurements of erythema and induration and assessment of other adverse events of pain/tenderness, bleeding, urticaria, infection, or blistering/ulcerating. Participants are counted if they had any measurable eythema or induration, or reported any of the other listed adverse events. Reactions were reported as present or absent, and were not graded for severity.
Time Frame: Up to 28 Days
Population: All participants who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | A1 - MLSA in Healthy Non-Exposed Participants | B1 - MLSA in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 5 | 45 | 20 | 20 | 20 | 20
Participants
  Erythema | 4 | 10 | 2 | 4 | 11 | 12
  Induration | 1 | 12 | 1 | 2 | 5 | 7
  Pain/Tenderness | 0 | 3 | 1 | 0 | 1 | 0
  Bleeding | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria | 0 | 0 | 0 | 0 | 0 | 1
  Infection | 0 | 0 | 0 | 0 | 0 | 1
  Blistering/Ulcerating | 0 | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Number of Participants With the Reaction of Itching to the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 1.0 Microgram
Description: as for outcome 2
Time Frame: Up to 28 Days
Population: All participants in Groups B and C who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | B1 - MLSA in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 45 | 20 | 20 | 20 | 20
Participants | 0 | 0 | 0 | 4 | 1

5. Primary Outcome: Number of Participants With Reactions to the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 0.1 Microgram
Description: as for outcome 3
Time Frame: Up to 28 Days
Population: All participants who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Groups:
- A2 - MLC in Healthy Non-Exposed Participants: 5 healthy non-exposed participants received 1.0 mcg of MLCwA, 0.1 mcg of M. leprae Cell Wall Antigen (MLCwA), 5 TU Purified Protein Derivative/Tubersol®, saline (NaCl)
Arm/Group | A2 - MLC in Healthy Non-Exposed Participants | B2 - MLC in Healthy Non-Exposed Participants | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 5 | 45 | 20 | 20 | 20 | 20
Participants
  Erythema | 0 | 1 | 1 | 8 | 5 | 5
  Induration | 0 | 1 | 0 | 5 | 5 | 3
  Pain/Tenderness | 0 | 0 | 0 | 0 | 0 | 0
  Bleeding | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria | 0 | 0 | 0 | 0 | 0 | 0
  Infection | 0 | 0 | 0 | 0 | 0 | 0
  Blistering/Ulcerating | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Reaction of Itching to the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 0.1 Microgram
Description: as for outcome 2
Time Frame: Up to 28 Days
Measure: Number; unit: Participants
Arm/Group | B2 - MLC in Healthy Non-Exposed Participants | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 45 | 20 | 20 | 20 | 20
Participants | 0 | 0 | 2 | 1 | 0

7. Primary Outcome: Number of Participants With Reactions to the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 1.0 Microgram
Description: as for outcome 3
Time Frame: Up to 28 Days
Population: All participants who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | A2 - MLC in Healthy Non-Exposed Participants | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 5 | 45 | 20 | 20 | 20 | 20
Participants
  Erythema | 3 | 11 | 2 | 5 | 8 | 14
  Induration | 1 | 10 | 0 | 3 | 9 | 9
  Pain/Tenderness | 0 | 0 | 1 | 1 | 1 | 2
  Bleeding | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria | 0 | 0 | 0 | 0 | 0 | 0
  Infection | 0 | 0 | 0 | 0 | 0 | 0
  Blistering/Ulcerating | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With the Reaction of Itching to the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 1.0 Microgram
Description: as for outcome 2
Time Frame: Up to 28 Days
Population: All participants in Groups B and C who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 45 | 20 | 20 | 20 | 20
Participants | 1 | 0 | 1 | 5 | 6

9. Primary Outcome: Number of Participants With Reactions to the Antigen Purified Protein Derivative (PPD)
Description: as for outcome 3
Time Frame: Up to 28 Days
Population: All participants who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | A1 - MLSA in Healthy Non-Exposed Participants | A2 - MLC in Healthy Non-Exposed Participants | B1 - MLSA in Healthy Non-Exposed Participants | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 5 | 5 | 45 | 45 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
Participants
  Erythema | 5 | 4 | 33 | 33 | 12 | 13 | 17 | 20 | 9 | 14 | 17 | 20
  Induration | 5 | 4 | 33 | 31 | 11 | 11 | 16 | 18 | 11 | 11 | 16 | 18
  Pain/Tenderness | 1 | 2 | 12 | 13 | 6 | 7 | 5 | 9 | 3 | 1 | 3 | 3
  Bleeding | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blistering/Ulcerating | 1 | 0 | 0 | 4 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0

10. Primary Outcome: Number of Participants With the Reaction of Itching to the Antigen Purified Protein Derivative (PPD)
Description: as for outcome 2
Time Frame: Up to 28 Days
Population: All participants in Groups B and C who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Groups:
- C1 - High Dose in BT/TT Leprosy Patients: 20 borderline tuberculoid/tuberculoid (BT/TT) leprosy patients received 1.0 mcg of MLSA-LAM, 1.0 mcg of MLCwA and 2TU Purified Protein Derivative/RT-23
Arm/Group | B1 - MLSA in Healthy Non-Exposed Participants | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 45 | 45 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
Participants | 17 | 17 | 5 | 5 | 9 | 14 | 0 | 8 | 5 | 12

11. Primary Outcome: Mean Diameter of Erythema at Site of Injection With the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 0.1 Micrograms
Description: If erythema was present, it was measured in millimeters for participants in Groups C1 and C1b only, who returned to the clinic at Days 3 and 7, and at Day 28 if reactions were still present.
Time Frame: Day 3
Population: The analysis population is restricted to participants in Group C1b who had measurable erythema at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 5 | 4 | 2
Millimeters | 12.6 (4.2) | 9.8 (1.8) | 9.3 (0.6)

12. Primary Outcome: Mean Diameter of Erythema at Site of Injection With the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 0.1 Micrograms
Description: as for outcome 11
Time Frame: Day 7
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 4 | 3 | 3
Millimeters | 11.3 (3.4) | 10.3 (0.8) | 9.8 (2.4)

13. Primary Outcome: Mean Diameter of Erythema at Site of Injection With the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 1.0 Micrograms
Description: as for outcome 11
Time Frame: Day 3
Population: The analysis population is restricted to participants in Group C1 who had measurable erythema at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 1 | 2 | 7 | 8
Millimeters | 20.0 | 23.3 (4.6) | 13.0 (5.9) | 14.8 (6.5)

14. Primary Outcome: Mean Diameter of Erythema at Site of Injection With the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 1.0 Micrograms
Description: as for outcome 11
Time Frame: Day 7
Population: The analysis population is restricted to participants in Group C1 who had measurable erythema at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 1 | 2 | 9 | 10
Millimeters | 16.0 | 20.3 (5.3) | 13.8 (6.6) | 14.3 (6.6)

15. Primary Outcome: Mean Diameter of Erythema at Site of Injection With the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 0.1 Micrograms
Description: as for outcome 11
Time Frame: Day 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 7 | 6 | 5
Millimeters | 15.1 (3.3) | 13.0 (4.6) | 9.6 (2.3)

16. Primary Outcome: Mean Diameter of Erythema at Site of Injection With the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 0.1 Micrograms
Description: as for outcome 11
Time Frame: Day 7
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 5 | 6 | 4
Millimeters | 12.1 (5.0) | 12.2 (3.4) | 8.9 (1.4)

17. Primary Outcome: Mean Diameter of Erythema at Site of Injection With the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 1.0 Micrograms
Description: as for outcome 11
Time Frame: Day 3
Population: The analysis population is restricted to participants in Group C1 who had measurable erythema at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 1 | 3 | 9 | 11
Millimeters | 9.0 | 20.8 (2.9) | 14.7 (5.7) | 15.0 (6.1)

18. Primary Outcome: Mean Diameter of Erythema at Site of Injection With the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 1.0 Micrograms
Description: as for outcome 11
Time Frame: Day 7
Population: The analysis population is restricted to participants in Group C1 who had measurable erythema at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 3 | 8 | 11
Millimeters | 17.8 (7.0) | 16.4 (5.1) | 13.8 (5.3)

19. Primary Outcome: Mean Diameter of Erythema at Site of Injection With the Antigen Purified Protein Derivative (PPD)
Description: as for outcome 11
Time Frame: Day 3
Population: The analysis population is restricted to participants in Group C1 and C1b who had measurable erythema at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 12 | 12 | 16 | 20 | 8 | 13 | 16 | 20
Millimeters | 20.4 (9.4) | 20.7 (8.0) | 19.3 (9.8) | 22.4 (7.1) | 18.1 (6.0) | 17.8 (4.8) | 17.6 (8.1) | 21.1 (7.0)

20. Primary Outcome: Mean Diameter of Erythema at Site of Injection With the Antigen Purified Protein Derivative (PPD)
Description: as for outcome 11
Time Frame: Day 7
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 9 | 12 | 16 | 20 | 10 | 12 | 17 | 20
Millimeters | 18.6 (5.4) | 19.0 (6.5) | 17.8 (5.7) | 20.9 (4.6) | 16.8 (4.2) | 17.1 (4.3) | 16.4 (6.2) | 19.1 (4.2)

21. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 0.1 Micrograms
Description: If induration was present, it was measured in millimeters at Days 2 (Group A), 3 (all groups) and 7 (Groups B and C), and at Day 28 if reactions were still present (all groups).
Time Frame: Day 3
Population: The analysis population is restricted to participants who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | B1 - MLSA in Healthy Non-Exposed Participants | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts
Number analyzed (Participants) | 2 | 4 | 2
Millimeters | 5.0 (3.5) | 14.0 (3.2) | 10.8 (1.1)

22. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 0.1 Micrograms
Description: as for outcome 21
Time Frame: Day 7
Population: The analysis population is restricted to participants in Groups B1 and C1b who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | B1 - MLSA in Healthy Non-Exposed Participants | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts
Number analyzed (Participants) | 1 | 4 | 3
Millimeters | 4.5 | 11.3 (3.4) | 10.3 (0.8)

23. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 1.0 Micrograms
Description: as for outcome 21
Time Frame: Day 2
Population: The analysis population is restricted to participants in Group A1 who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | A1 - MLSA in Healthy Non-Exposed Participants
Number analyzed (Participants) | 1
Millimeters | 25.0

24. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 1.0 Micrograms
Description: as for outcome 21
Time Frame: Day 3
Population: The analysis population is restricted to participants in Groups A1, B1 and C1 who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | A1 - MLSA in Healthy Non-Exposed Participants | B1 - MLSA in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 1 | 9 | 1 | 2 | 5 | 7
Millimeters | 20.0 | 9.4 (5.5) | 20.0 | 21.3 (2.5) | 14.4 (6.5) | 14.1 (4.7)

25. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen Mycobacterium (M.) Leprae Soluble Antigen (MLSA)-Lipoarabinomannan (LAM) at Doses of 1.0 Micrograms
Description: as for outcome 21
Time Frame: Day 7
Population: The analysis population is restricted to participants in Groups B1 and C1 who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | B1 - MLSA in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 12 | 1 | 2 | 5 | 7
Millimeters | 8.1 (3.4) | 16 | 16.3 (9.5) | 17.1 (6.2) | 6.4 (2.9)

26. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 0.1 Micrograms
Description: as for outcome 21
Time Frame: Day 3
Population: The analysis population is restricted to participants in Groups A2, B2 and C1b who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 5 | 4 | 3
Millimeters | 14.8 (4) | 11.5 (5.1) | 8.3 (2.1)

27. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 0.1 Micrograms
Description: as for outcome 21
Time Frame: Day 7
Population: The analysis population is restricted to participants in Groups B2 and C1b who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | B2 - MLC in Healthy Non-Exposed Participants | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 1 | 5 | 5 | 1
Millimeters | 7.0 | 11.4 (4.0) | 11.8 (3.7) | 10.0

28. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 1.0 Micrograms
Description: as for outcome 21
Time Frame: Day 2
Population: The analysis population is restricted to participants in Group A2 who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | A2 - MLC in Healthy Non-Exposed Participants
Number analyzed (Participants) | 1
Millimeters | 25.0

29. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 1.0 Micrograms
Description: as for outcome 21
Time Frame: Day 3
Population: The analysis population is restricted to participants in Groups A2, B2 and C1 who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | A2 - MLC in Healthy Non-Exposed Participants | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 1 | 7 | 3 | 9 | 9
Millimeters | 16.5 | 9.8 (5.1) | 20.1 (1.3) | 14.2 (4.9) | 14.6 (5.4)

30. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen M. Leprae Cell Wall Antigen (MLCwA) at Doses of 1.0 Micrograms
Description: as for outcome 21
Time Frame: Day 7
Population: The analysis population is restricted to participants in Groups B2 and C1 who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 10 | 1 | 8 | 7
Millimeters | 9.0 (4.7) | 23.5 | 13.8 (7.5) | 10.2 (4.9)

31. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen Purified Protein Derivative (PPD)
Description: as for outcome 21
Time Frame: Day 2
Population: The analysis population is restricted to participants in Groups A1 and A2 who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | A1 - MLSA in Healthy Non-Exposed Participants | A2 - MLC in Healthy Non-Exposed Participants
Number analyzed (Participants) | 5 | 4
Millimeters | 19.3 (15.2) | 25.5 (11.0)

32. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen Purified Protein Derivative (PPD)
Description: as for outcome 21
Time Frame: Day 3
Population: The analysis population is restricted to participants in all groups who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | A1 - MLSA in Healthy Non-Exposed Participants | A2 - MLC in Healthy Non-Exposed Participants | B1 - MLSA in Healthy Non-Exposed Participants | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 5 | 4 | 30 | 29 | 11 | 11 | 16 | 18 | 11 | 11 | 16 | 18
Millimeters | 19.1 (9.7) | 20.5 (8.2) | 15.1 (5.6) | 18.8 (6.5) | 18.7 (6.3) | 21 (5.4) | 17.2 (6.0) | 20.1 (4.6) | 18.8 (6.3) | 21.0 (5.4) | 17.2 (6.0) | 20.1 (4.6)

33. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen Purified Protein Derivative (PPD)
Description: as for outcome 21
Time Frame: Day 7
Population: The analysis population is restricted to participants in Groups B1, B2, C1 and C1b who had measurable induration at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | B1 - MLSA in Healthy Non-Exposed Participants | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 33 | 31 | 8 | 11 | 15 | 18 | 8 | 11 | 15 | 18
Millimeters | 14.0 (5.7) | 16.0 (5.6) | 18.3 (5.8) | 18.8 (6.8) | 17.0 (5.6) | 17.5 (5.6) | 18.3 (5.8) | 18.8 (6.8) | 17.0 (5.6) | 17.5 (5.6)

34. Primary Outcome: Mean Diameter of Induration at Site of Injection With the Antigen Purified Protein Derivative (PPD)
Description: as for outcome 21
Time Frame: Day 28
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | A1 - MLSA in Healthy Non-Exposed Participants | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | C1b - Low Dose MLSA and MLC in Healthy Contacts
Number analyzed (Participants) | 1 | 4 | 1 | 1
Millimeters | 16.0 | 13.5 (0) | 8.0 | 8

35. Primary Outcome: Number of Participants With QuantiFERON Responses Based on the Presence or Absence of Induration at the Injection Site for the Antigen MLSA-LAM at Doses of 0.1 Microgram.
Description: Blood collection for the QuantiFERON assessment was at Day 0 prior to antigen administration. Participants are considered to have a positive QuantiFERON response if the result was greater than 0. The categories present the number of participants who are positive or negative by QuantiFERON based on whether or not induration was assessed as present at any of the follow up visit assessments. A fifth category is listed to report the number of participants who were missing either a QuantiFERON result or induration assessment. The categories are mutually exclusive.
Time Frame: Day 0 for QuantiFERON; Days 3, 7, and 28 for induration
Population: All evaluable participants in Group C1b who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 19 | 20 | 20 | 20
Participants
  Positive QuantiFERON and Induration > 0 mm | 0 | 5 | 3 | 1
  Negative QuantiFERON and Induration = 0 mm | 2 | 1 | 0 | 1
  Negative QuantiFERON and Induration > 0 mm | 0 | 0 | 0 | 0
  Positive QuantiFERON and Induration = 0 mm | 17 | 12 | 14 | 15
  Missing QuantiFERON result and/or Induration | 0 | 2 | 3 | 3

36. Primary Outcome: Number of Participants With QuantiFERON Responses Based on the Presence or Absence of Induration at the Injection Site for the Antigen MLSA-LAM at Doses of 1.0 Microgram.
Description: as for outcome 35
Time Frame: Day 0 for QuantiFERON; Days 3, 7, and 28 for induration
Population: All participants in Group C1 who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants
  Positive QuantiFERON and Induration > 0 mm | 4 | 5 | 2 | 0
  Negative QuantiFERON and Induration = 0 mm | 5 | 10 | 9 | 12
  Negative QuantiFERON and Induration > 0 mm | 2 | 4 | 0 | 1
  Positive QuantiFERON and Induration = 0 mm | 9 | 1 | 9 | 7
  Missing QuantiFERON result and/or Induration | 0 | 0 | 0 | 0

37. Primary Outcome: Number of Participants With QuantiFERON Responses Based on the Presence or Absence of Induration at the Injection Site for the Antigen MLCwA at Doses of 0.1 Microgram.
Description: as for outcome 35
Time Frame: Day 0 for QuantiFERON; Days 3, 7, and 28 for induration
Population: All evaluable participants in Group C1b who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 19 | 20 | 20 | 20
Participants
  Positive QuantiFERON and Induration > 0 mm | 0 | 6 | 5 | 3
  Negative QuantiFERON and Induration = 0 mm | 3 | 1 | 0 | 1
  Negative QuantiFERON and Induration > 0 mm | 0 | 0 | 0 | 0
  Positive QuantiFERON and Induration = 0 mm | 16 | 11 | 12 | 13
  Missing QuantiFERON result and/or Induration | 0 | 2 | 3 | 3

38. Primary Outcome: Number of Participants With QuantiFERON Responses Based on the Presence or Absence of Induration at the Injection Site for the Antigen MLCwA at Doses of 1.0 Microgram.
Description: as for outcome 35
Time Frame: Day 0 for QuantiFERON; Days 3, 7, and 28 for induration
Population: All participants in Group C1 who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants
  Positive QuantiFERON and Induration > 0 mm | 0 | 2 | 8 | 4
  Negative QuantiFERON and Induration = 0 mm | 9 | 10 | 3 | 7
  Negative QuantiFERON and Induration > 0 mm | 0 | 1 | 2 | 6
  Positive QuantiFERON and Induration = 0 mm | 11 | 7 | 7 | 3
  Missing QuantiFERON result and/or Induration | 0 | 0 | 0 | 0

39. Primary Outcome: Number of Participants With QuantiFERON Responses Based on the Presence or Absence of Induration at the Injection Site for the Antigen PPD.
Description: as for outcome 35
Time Frame: Day 0 for QuantiFERON; Days 3, 7, and 28 for induration
Population: All evaluable participants in Groups C1 and C1b who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 19 | 20 | 20 | 20
Participants
  Positive QuantiFERON and Induration > 0 mm | 10 | 11 | 15 | 17 | 9 | 13 | 14 | 17
  Negative QuantiFERON and Induration = 0 mm | 4 | 3 | 0 | 1 | 2 | 0 | 0 | 0
  Negative QuantiFERON and Induration > 0 mm | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
  Positive QuantiFERON and Induration = 0 mm | 5 | 5 | 3 | 1 | 8 | 5 | 3 | 0
  Missing QuantiFERON result and/or Induration | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3

40. Primary Outcome: Number of Participants Positive for Phenolic Glycolipid-1 (PGL-1) by QuantiFERON Results and the Presence or Absence of Induration at the Injection Site for the Antigen MLSA-LAM at Doses of 0.1 Microgram
Description: Blood was collected at Day 0 prior to antigen administration for the assessment of PGL-1 and QuantiFERON. The mutually exclusive categories present the number of participants positive or negative by the two assays based on presence of induration at any of the follow up visit assessments. Results for PGL-1 of weakly, moderately or strongly positive are grouped as positive. A result greater than 0 is considered positive for QuantiFERON. A fifth category is listed to report the number of participants who were missing either assay result or the induration assessment.
Time Frame: Day 0 for PGL-1 and QuantiFERON; Days 3, 7, and 28 for induration
Population: All evaluable participants in Group C1b who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 19 | 20 | 20 | 20
Participants
  Pos PGL, Neg QuantiFERON and Induration = 0 mm | 1 | 0 | 0 | 0
  Neg PGL, Pos QuantiFERON and Induration > 0 mm | 0 | 3 | 3 | 0
  Pos PGL, Pos QuantiFERON and Induration > 0 mm | 0 | 2 | 0 | 1
  Neg PGL, Neg QuantiFERON and Induration = 0 mm | 1 | 1 | 0 | 1
  Neg PGL, Neg QuantiFERON and Induration = 0 mm | 0 | 0 | 0 | 0
  Pos PGL, Neg QuantiFERON and Induration > 0 mm | 0 | 0 | 0 | 0
  Neg PGL, Pos QuantiFERON and Induration > 0 mm | 4 | 6 | 11 | 13
  Pos PGL, Pos QuantiFERON and Induration = 0 mm | 13 | 6 | 3 | 2
  Missing Either Assay Result or Induration | 0 | 2 | 3 | 3

41. Primary Outcome: Number of Participants Positive for Phenolic Glycolipid-1 (PGL-1) by QuantiFERON Results and the Presence or Absence of Induration at the Injection Site for the Antigen MLSA-LAM at Doses of 1.0 Microgram
Description: as for outcome 40
Time Frame: Day 0 for PGL-1 and QuantiFERON; Days 3, 7, and 28 for induration
Population: All participants in Group C1 who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants
  Pos PGL, Neg QuantiFERON and Induration = 0 mm | 3 | 10 | 6 | 12
  Neg PGL, Pos QuantiFERON and Induration > 0 mm | 2 | 1 | 0 | 0
  Pos PGL, Pos QuantiFERON and Induration > 0 mm | 2 | 4 | 2 | 0
  Neg PGL, Neg QuantiFERON and Induration = 0 mm | 2 | 0 | 2 | 0
  Neg PGL, Neg QuantiFERON and Induration = 0 mm | 0 | 2 | 0 | 0
  Pos PGL, Neg QuantiFERON and Induration > 0 mm | 2 | 2 | 0 | 1
  Neg PGL, Pos QuantiFERON and Induration > 0 mm | 4 | 0 | 5 | 0
  Pos PGL, Pos QuantiFERON and Induration = 0 mm | 5 | 1 | 4 | 7
  Missing Either Assay Result or Induration | 0 | 0 | 1 | 0

42. Primary Outcome: Number of Participants Positive for Phenolic Glycolipid-1 (PGL-1) by QuantiFERON Results and the Presence or Absence of Induration at the Injection Site for the Antigen MLCwA at Doses of 0.1 Microgram
Description: as for outcome 40
Time Frame: Day 0 for PGL-1 and QuantiFERON; Days 3, 7, and 28 for induration
Population: All evaluable participants in Group C1b who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 19 | 20 | 20 | 20
Participants
  Pos PGL, Neg QuantiFERON and Induration = 0 mm | 2 | 0 | 0 | 0
  Neg PGL, Pos QuantiFERON and Induration > 0 mm | 0 | 4 | 5 | 2
  Pos PGL, Pos QuantiFERON and Induration > 0 mm | 0 | 2 | 0 | 1
  Neg PGL, Neg QuantiFERON and Induration = 0 mm | 1 | 1 | 0 | 1
  Neg PGL, Neg QuantiFERON and Induration = 0 mm | 0 | 0 | 0 | 0
  Pos PGL, Neg QuantiFERON and Induration > 0 mm | 0 | 0 | 0 | 0
  Neg PGL, Pos QuantiFERON and Induration > 0 mm | 4 | 5 | 9 | 11
  Pos PGL, Pos QuantiFERON and Induration = 0 mm | 12 | 6 | 3 | 2
  Missing Either Assay Result or Induration | 0 | 2 | 3 | 3

43. Primary Outcome: Number of Participants Positive for Phenolic Glycolipid-1 (PGL-1) by QuantiFERON Results and the Presence or Absence of Induration at the Injection Site for the Antigen MLCwA at Doses of 1.0 Microgram
Description: as for outcome 40
Time Frame: Day 0 for PGL-1 and QuantiFERON; Days 3, 7, and 28 for induration
Population: All participants in Group C1 who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants
  Pos PGL, Neg QuantiFERON and Induration = 0 mm | 9 | 7 | 1 | 6
  Neg PGL, Pos QuantiFERON and Induration > 0 mm | 0 | 0 | 5 | 1
  Pos PGL, Pos QuantiFERON and Induration > 0 mm | 0 | 2 | 3 | 3
  Neg PGL, Neg QuantiFERON and Induration = 0 mm | 0 | 3 | 2 | 1
  Neg PGL, Neg QuantiFERON and Induration = 0 mm | 0 | 0 | 0 | 1
  Pos PGL, Neg QuantiFERON and Induration > 0 mm | 0 | 0 | 2 | 5
  Neg PGL, Pos QuantiFERON and Induration > 0 mm | 0 | 4 | 1 | 0
  Pos PGL, Pos QuantiFERON and Induration = 0 mm | 11 | 3 | 6 | 3
  Missing Either Assay Result or Induration | 0 | 1 | 0 | 0

44. Primary Outcome: Number of Participants Positive for Phenolic Glycolipid-1 (PGL-1) by QuantiFERON Results and the Presence or Absence of Induration at the Injection Site for the Antigen PPD
Description: as for outcome 40
Time Frame: Day 0 for PGL-1 and QuantiFERON; Days 3, 7, and 28 for induration
Population: All evaluable participants in Group C1 and C1b who received the antigen are included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 19 | 20 | 20 | 20
Participants
  Pos PGL, Neg QuantiFERON and Induration = 0 mm | 4 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Neg PGL, Pos QuantiFERON and Induration > 0 mm | 0 | 4 | 5 | 3 | 2 | 6 | 12 | 14
  Pos PGL, Pos QuantiFERON and Induration > 0 mm | 10 | 7 | 10 | 14 | 7 | 7 | 2 | 3
  Neg PGL, Neg QuantiFERON and Induration = 0 mm | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  Neg PGL, Neg QuantiFERON and Induration = 0 mm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pos PGL, Neg QuantiFERON and Induration > 0 mm | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
  Neg PGL, Pos QuantiFERON and Induration > 0 mm | 0 | 1 | 3 | 0 | 2 | 4 | 2 | 0
  Pos PGL, Pos QuantiFERON and Induration = 0 mm | 5 | 4 | 0 | 1 | 6 | 1 | 1 | 0
  Missing Either Assay Result or Induration | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 3

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events were collected for the duration of the participant's participation in the study, up to 28 days after study product administration.
Description: Solicited reactions were assessed by clinic staff at Days 0, 3, and 7, and at Day 28 if reactions were present at Day 7. Participants are counting as having the reaction if present at any of these days. Events are counted separately for the solicited reactions at each injection site.
Arm/Group | A1 - MLSA in Healthy Non-Exposed Participants | A2 - MLC in Healthy Non-Exposed Participants | B1 - MLSA in Healthy Non-Exposed Participants | B2 - MLC in Healthy Non-Exposed Participants | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts | CI - High Dose MLSA and MLC in TB Patients | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients | C1b - Low Dose MLSA and MLC in Healthy Contacts | C1b - Low Dose MLSA and MLC in TB Patients
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 2/45 | 0/45 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/5 | 4/5 | 36/45 | 35/45 | 13/20 | 15/20 | 19/20 | 20/20 | 11/20 | 16/20 | 18/20 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1 - MLSA in Healthy Non-Exposed Participants (N=5) | A2 - MLC in Healthy Non-Exposed Participants (N=5) | B1 - MLSA in Healthy Non-Exposed Participants (N=45) | B2 - MLC in Healthy Non-Exposed Participants (N=45) | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients (N=20) | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients (N=20) | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts (N=20) | CI - High Dose MLSA and MLC in TB Patients (N=20) | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients (N=20) | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients (N=20) | C1b - Low Dose MLSA and MLC in Healthy Contacts (N=20) | C1b - Low Dose MLSA and MLC in TB Patients (N=20)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1 - MLSA in Healthy Non-Exposed Participants (N=5) | A2 - MLC in Healthy Non-Exposed Participants (N=5) | B1 - MLSA in Healthy Non-Exposed Participants (N=45) | B2 - MLC in Healthy Non-Exposed Participants (N=45) | C1 - High Dose MLSA and MLC in BL/LL Leprosy Patients (N=20) | C1 - High Dose MLSA and MLC in BT/TT Leprosy Patients (N=20) | C1 - High Dose MLSA and MLC in BL/LL Healthy Contacts (N=20) | CI - High Dose MLSA and MLC in TB Patients (N=20) | C1b - Low Dose MLSA and MLC in BL/LL Leprosy Patients (N=20) | C1b - Low Dose MLSA and MLC in BT/TT Leprosy Patients (N=20) | C1b - Low Dose MLSA and MLC in Healthy Contacts (N=20) | C1b - Low Dose MLSA and MLC in TB Patients (N=20)
Erythema (Skin and subcutaneous tissue disorders) | 5 (9) | 4 (7) | 36 (46) | 34 (45) | 13 (16) | 15 (22) | 19 (36) | 20 (46) | 11 (11) | 16 (27) | 18 (26) | 20 (27)
Induration (General disorders) | 5 (6) | 4 (5) | 34 (46) | 31 (42) | 12 (12) | 14 (16) | 18 (30) | 18 (34) | 9 (11) | 15 (20) | 17 (22) | 20 (21)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 17 (17) | 17 (18) | 5 (5) | 6 (6) | 10 (25) | 15 (21) | 0 (0) | 9 (11) | 6 (7) | 12 (12)
Pain (General disorders) | 1 (1) | 2 (2) | 14 (16) | 13 (13) | 7 (8) | 8 (8) | 5 (7) | 9 (11) | 3 (3) | 1 (1) | 4 (4) | 3 (3)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Type IV hypersensitivity reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less